CLINICAL TRIAL: NCT03112499
Title: The Effect of Three Endourological Procedures for the Management of Renal Calculi Regarding Acute Kidney Injury: a Prospective Randomized 3-arm Study.
Brief Title: The Effect of Three Endourological Procedures for the Management of Renal Calculi Regarding Acute Kidney Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for the Study of Urological Diseases, Greece (Other)
Responsible Party: Principal Investigator, Dimitrios Hatzichristou, President, Institute for the Study of Urological Diseases, Greece
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1343/2017
Record Dates: First submitted 2017-03-28; First posted 2017-04-13 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Renal Calculi; Renal Insufficiency
Keywords: Acute Kidney Injury; PCNL; mini-PCNL; RIRS; urine biomarkers
MeSH Terms: conditions — Kidney Calculi; Renal Insufficiency; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PCNL Group (Active Comparator): Patients with renal calculi 10-30mm in maximal diameter in who percutaneous nephrolithotomy (PCNL) will be conducted
  Interventions: Procedure: PCNL
- mini-PCNL Group (Active Comparator): Patients with renal calculi 10-30mm in maximal diameter in who mini- percutaneous nephrolithotomy (mini-PCNL) will be conducted
  Interventions: Procedure: mini-PCNL
- RIRS Group (Active Comparator): Patients with renal calculi 10-30mm in maximal diameter in who retrograde intrarenal surgery (RIRS) will be conducted
  Interventions: Procedure: RIRS

INTERVENTIONS:
Procedure: PCNL — Under general anesthesia and patient in prone position, with the use of a flexible cystoscope an open-ended ureteral catheter 5F / 70cm is positioned to the proximal ureter. Retrograde pyelography is performed and the most appropriate calyx is accessed with the use of ultrasound, under fluoroscopic guidance. A 0.035 guide wire is inserted into the ureter and then replaced with an extra stiff wire. Using either balloon (20 atm) or Amplatz serial dilators a 30F access channel is created. Lithotripsy is performed using ultrasound lithotripter and stone fragments are removed by grasping forceps. At the end of the operation a 18F Council type catheter is placed into the kidney for drainage of urine and an indwelling JJ catheter is inserted in the ipsilateral ureter. Council and JJ catheter are removed,in the absence of complications, the second and tenth postoperative day, respectively.
  Arms: PCNL Group
Procedure: mini-PCNL — Under general anesthesia and patient in prone position, with the use of a flexible cystoscope an open-ended ureteral catheter 5F / 70cm is positioned to the proximal ureter. Retrograde pyelography is performed and the most appropriate calyx is accessed with the use of ultrasound, under fluoroscopic guidance. A 0.035 guide wire is inserted into the ureter and then replaced with an extra stiff wire. Using Amplatz serial dilators a 16F access channel is created. Lithotripsy is performed using using 270mm Ho: YAG laser fiber and stone fragments are removed by grasping forceps. At the end of the operation a 10F nephrostomy tube is placed into the kidney for drainage of urine and an indwelling JJ catheter is inserted in the ipsilateral ureter. Nephrostomy tube and JJ catheter are removed, in the absence of complications, the second and tenth postoperative day, respectively.
  Arms: mini-PCNL Group
Procedure: RIRS — Under general anesthesia and patient in lithotomy position, a 0.035 hydrophilic safety wire is inserted in the ureter under fluoroscopic guidance. Subsequently 8-10 F dilators are used for dilation of the ureter.Insertion of a second working wire follows above which a 14F ureteral sheath is placed. Lithotripsy with a flexible ureteroscope using 270mm Ho: YAG laser fiber follows.Remaining stone fragments are removed by a 2,2F nitinol basket. At the end of the operation a JJ indwelling ureteral catheter is placed over the safety wire. Discharge is performed in the absence of complications, the first postoperative day while JJ catheter is removed on the 10th postoperative day.
  Arms: RIRS Group

SUMMARY:
The main aim of the study is to investigate and compare the possible acute effect of standard PCNL, mini-PCNL and RIRS on renal function. Secondary aims are to investigate the efficacy (stone-free rate), safety (complication rate, long-term kidney function) and other parameters (operation, fluoroscopy and hospitalization time) concerning the 3 endourological operations (PCNL, mini- PCNL, RIRS) for the treatment of renal calculi.

DETAILED DESCRIPTION:
This is a 3-arm parallel group prospective randomized active-treatment clinical study. A total of 75 patients with renal calculi 10-30 mm in maximal diameter measured in abdominal CT scan will be recruited in this research protocol. Patient enrollment will be performed from patients referred to Urolithiasis Unit of the 1st Urology Department, G. Gennimatas Hospital, Aristotle University of Thessaloniki. In all potentially eligible patients full medical history, as well as demographic characteristics and drug treatment will be recorded, followed by a detailed physical examination and standard laboratory tests.

Eligible patients will be randomized to receive one of the following endourological techniques of nephrolithotripsy: standard PCNL, mini- PCNL or RIRS. All eligible patients will be randomised to one of the 3 groups, consisting of 25 patients, with an equal allocation ratio (1:1). The randomization sequence will be computer generated by the study coordinating team.

The primary and secondary measurements of the study will be carried in prespecified time-points that are listed below:

Point 0(P0): Screening visit:

Potentially eligible patients will be asked to provide written informed consent. We will record full medical history, concomitant medication, clinical examination, demographic characteristics, body weight, height, body mass index (BMI).

Point 1(P1): 1st day of hospitalization (Monday or Thursday):

Admission of the patient to the hospital where a routine preoperative control is conducted including: routine hematological and biochemical laboratory parameters (Hct, Hb, WBC, PLT, fasting glucose, urea, creatinine, serum electrolytes, SGOT, SGPT), chest X-ray and anesthesiological preoperative evaluation. Patient is randomized to be treated with one of the 3 endourological operations.

Point 2(P2): Operation day (Tuesday or Friday), 2 hours before the operation:

Urine sample is collected for measurement of urine biomarkers (NGAL, KIM-1, IL-18) and creatinine (baseline values). Blood sample is collected for creatinine measurement and eGFR is calculated.

Point 3(P3): Operation (PCNL, mini-PCNL or RIRS):

Operation, fluoroscopy time and intraoperative complications are recorded

Point 4(P4): 2 hours after the operation:

Urine sample is collected for measurement of urine biomarkers (NGAL, KIM-1, IL-18) and creatinine. Blood sample is collected for creatinine measurement and eGFR is calculated. A VAS pain score is completed. Urine output is measured. Postoperative complications are recorded.

Point 5(P5): 6 hours after the operation:

Urine sample is collected for measurement of urine biomarkers (NGAL, KIM-1, IL-18) and creatinine. Blood sample is collected for creatinine measurement and eGFR is calculated. A VAS pain score is completed. Urine output is measured. Postoperative complications are recorded.

Point 6(P6): 24 hours after the operation:

Urine sample is collected for measurement of urine biomarkers (NGAL, KIM-1, IL-18) and creatinine. Blood sample is collected for creatinine measurement and eGFR is calculated. A VAS pain score is completed. Urine output is measured. Postoperative complications are recorded.

Point 7(P7): 48 hours after the operation:

Urine sample is collected for measurement of urine biomarkers (NGAL, KIM-1, IL-18) and creatinine. Blood sample is collected for creatinine measurement and eGFR is calculated. A VAS pain score is completed. Urine output is measured. Potential postoperative complications are recorded.

Point 8(P8): 1 month after the operation:

CT scan is conducted for confirmation of treatment success and stone free status or not. Blood sample is collected for creatinine measurement and eGFR is calculated. Potential postoperative complications are recorded.

Point9(P9): 3 months after the operation:

Blood sample is collected for creatinine measurement and eGFR is calculated. Potential postoperative complications are recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged > 18 years old
2. Patients with renal stone or stones of 10-30 mm in maximal diameter measured in computed tomography scan.
3. Decision of the patient to receive surgical treatment
4. Ability to understand and provide a written informed consent to participate in the study.

Exclusion Criteria:

1. Solitary kidney (functional or organic)
2. Ureteral stone in the same system causing obstruction
3. Malignant tumor in the treated kidney
4. Stone in diverticulum
5. Diabetes or coronary heart disease.
6. History of surgery in the treated kidney
7. Recent intake of drugs that affect renal function or intravenous contrast agent
8. Concomitant urinary infection
9. Congenital anomalies of the urinary tract
10. Patients of whom incomplete clinical data or incomplete samples are available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
The change in urine NGAL/Cr value | 2 hours preoperative and 2 hours postoperatively
  Urine NGAL/Cr value in all patients undergone nephrolithotripsy with PCNL, mini-PCNL or RIRS technique will be measured using Elisa technique.

SECONDARY OUTCOMES:
The change in urine NGAL/Cr value | 2 hours preoperative and 6, 24, 48 hours postoperatively
  Urine NGAL/Cr value in all patients undergone nephrolithotripsy with PCNL, mini-PCNL or RIRS technique will be measured using Elisa technique.
The change in urine KIM-1/Cr value | 2 hours preoperative and 2, 6, 24, 48 hours postoperatively
  Urine KIM-1/Cr value in all patients undergone nephrolithotripsy with PCNL, mini-PCNL or RIRS technique will be measured using Elisa technique.
The change in urine IL-18/Cr value | 2 hours preoperative and 2, 6, 24, 48 hours postoperatively
  Urine IL-18/Cr value in all patients undergone nephrolithotripsy with PCNL, mini-PCNL or RIRS technique will be measured using Elisa technique.
The difference in the values of urine NGAL/Cr, KIM1/Cr and IL-18/Cr between the patients undergone nephrolithotripsy with standard PCNL and those undergone nephrolithotripsy with mini - PCNL technique | 2, 6, 24, 48 hours postoperatively
  Urine NGAL/Cr, KIM1/Cr and IL-18/Cr values in all patients undergone nephrolithotripsy with standard PCNL or mini-PCNL technique will be measured using Elisa technique.
The difference in the values of urine NGAL/Cr, KIM1/Cr and IL-18/Cr between the patients undergone nephrolithotripsy with standard PCNL and those undergone nephrolithotripsy with RIRS technique | 2, 6, 24, 48 hours postoperatively
  Urine NGAL/Cr, KIM1/Cr and IL-18/Cr values in all patients undergone nephrolithotripsy with standard PCNL or RIRS technique will be measured using Elisa technique.
The difference in the values of urine NGAL/Cr, KIM1/Cr and IL-18/Cr between the patients undergone nephrolithotripsy with mini -PCNL and those undergone nephrolithotripsy with RIRS technique | 2, 6, 24, 48 hours postoperatively
  Urine NGAL/Cr, KIM1/Cr and IL-18/Cr values in all patients undergone nephrolithotripsy with mini-PCNL or RIRS technique will be measured using Elisa technique.
The presence of Acute Kidney Injury(AKI) in patients undergoing PCNL, mini-PCNL or RIRS | from the time of operation until 48 hours postoperatively
  Potential presence of AKI in patients undergoing PCNL or mini-PCNL or RIRS for the treatment of renal stones of 10-30mm in maximal diameter according to the KDIGO criteria, defined as: Serum Cr rise of 0,3mg/dl (≥26μmol/L) within 48 hours or 50-99% Cr rise from baseline within 7 days (1, 50-1, 99 x baseline) or urine output <0, 5/kg/h for more than 6 hours
The change in serum creatinine and eGFR values postoperatively in all patients undergone nephrolithotripsy with PCNL, mini-PCNL or RIRS technique. | 1 month and 3 months postoperatively
  * Serum creatinine levels will be measured using autoanalyzer
  * Calculation of eGFR will be done according to the equation CKD-EPI:
  GFR = 141 * min(Scr/κ,1)α * max(Scr/κ, 1)-1.209 * 0.993Age * 1.018 [if female] * 1.159 [if black]
  *Scr is serum creatinine (mg/dL), κ is 0.7 for females and 0.9 for males, α is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/κ or 1, and max indicates the maximum of Scr/κ or 1
Percent of patients achieving treatment success and stone-free state in after undergone nephrolithotripsy with PCNL, mini-PCNL or RIRS technique. | 4 weeks postoperatively
  * Treatments success (considered as absence of any stone or presence of residual stone fragment 4mm)
  * Stone-free rate (considered as absence of any stone) in CT scan
Overall complications rates in all patients undergone nephrolithotripsy with PCNL, mini-PCNL or RIRS technique. | from the time of operation until the 3 month follow up visit
  Complications will be recorded according the Clavien Dindo grading system
Operation time in all patients undergone nephrolithotripsy with PCNL, mini-PCNL or RIRS technique. | - from the renal puncture until the placement of the renal tube in the end of the PCNL or mini-PCNL operations/- From the insertion of the resectoscope into the bladder until the placement of the urethra catheter in the end of the RIRS operation
  Operation time will be recorded in minutes
Fluoroscopy time in all patients undergone nephrolithotripsy with PCNL, mini-PCNL or RIRS technique. | from the renal puncture until the placement of the renal tube in the end of the PCNL or mini-PCNL operations/- From the insertion of the resectoscope into the bladder until the placement of the urethra catheter in the end of the RIRS operation
  Fluoroscopy time will be recorded in minutes automatically by the fluoroscopic machine
Hospital stay duration in all patients undergone nephrolithotripsy with PCNL, mini-PCNL or RIRS technique. | From the day of operation until the day of discharge, up to 7 days
  Hospitalization time will be recorded in days
Postoperative pain, in all patients undergone nephrolithotripsy with PCNL, mini-PCNL or RIRS technique. | Immediately after the operation and in 2, 6, 24, 48 hours postoperatively.
  Postoperative pain will be measured by a visual analog scale (VAS) pain score

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Hatzichristou, Prof., Principal Investigator — Institute for the Study of Urological Diseases (ISUD)
Locations (1):
- G.Gennimatas Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Background] Haase M, Bellomo R, Devarajan P, Schlattmann P, Haase-Fielitz A; NGAL Meta-analysis Investigator Group. Accuracy of neutrophil gelatinase-associated lipocalin (NGAL) in diagnosis and prognosis in acute kidney injury: a systematic review and meta-analysis. Am J Kidney Dis. 2009 Dec;54(6):1012-24. doi: 10.1053/j.ajkd.2009.07.020. Epub 2009 Oct 21. PMID 19850388
- [Background] Vaidya VS, Waikar SS, Ferguson MA, Collings FB, Sunderland K, Gioules C, Bradwin G, Matsouaka R, Betensky RA, Curhan GC, Bonventre JV. Urinary biomarkers for sensitive and specific detection of acute kidney injury in humans. Clin Transl Sci. 2008 Dec;1(3):200-8. doi: 10.1111/j.1752-8062.2008.00053.x. PMID 19212447
- [Background] Lin X, Yuan J, Zhao Y, Zha Y. Urine interleukin-18 in prediction of acute kidney injury: a systemic review and meta-analysis. J Nephrol. 2015 Feb;28(1):7-16. doi: 10.1007/s40620-014-0113-9. Epub 2014 Jun 5. PMID 24899123
- [Background] Dede O, Dagguli M, Utangac M, Yuksel H, Bodakci MN, Hatipoglu NK, Sancaktutar AA, Penbegul N. Urinary expression of acute kidney injury biomarkers in patients after RIRS: it is a prospective, controlled study. Int J Clin Exp Med. 2015 May 15;8(5):8147-52. eCollection 2015. PMID 26221383
- [Background] Daggulli M, Utangac MM, Dede O, Bodakci MN, Hatipoglu NK, Penbegul N, Sancaktutar AA, Bozkurt Y, Soylemez H. Potential biomarkers for the early detection of acute kidney injury after percutaneous nephrolithotripsy. Ren Fail. 2016;38(1):151-6. doi: 10.3109/0886022X.2015.1073494. Epub 2015 Oct 19. PMID 26481764
- [Background] Balasar M, Piskin MM, Topcu C, Demir LS, Gurbilek M, Kandemir A, Ozturk A. Urinary kidney injury molecule-1 levels in renal stone patients. World J Urol. 2016 Sep;34(9):1311-6. doi: 10.1007/s00345-016-1765-y. Epub 2016 Jan 21. PMID 26795762
- [Derived] Soderberg L, Ergun O, Ding M, Parker R, Borofsky MS, Pais V, Dahm P. Percutaneous nephrolithotomy versus retrograde intrarenal surgery for treatment of renal stones in adults. Cochrane Database Syst Rev. 2023 Nov 13;11(11):CD013445. doi: 10.1002/14651858.CD013445.pub2. PMID 37955353